CLINICAL TRIAL: NCT02333903
Title: Effects of an Adapted Physical Activity Program on Health and Physical Condition After Sleeve Gastrectomy
Brief Title: Adapted Physical Activity Program After Sleeve Gastrectomy
Acronym: PEEPSO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Université de Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-P0030
Record Dates: First submitted 2014-12-29; First posted 2015-01-07 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-01

CONDITIONS: Obesity
Keywords: Obesity; Sleeve gastrectomy; Personalized physical activity program; Body Composition; Fat mass; Lean mass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Personalized Physical Activity (Experimental): Patients will undergo a personalized physical activity program after sleeve gastrectomy.
  Interventions: Other: Personalized Physical Activity
- Regular Activity (No Intervention): Patients will have regular physical activity after sleeve gastrectomy.

INTERVENTIONS:
Other: Personalized Physical Activity — 1.5 hours physical training sessions, twice a week for 1 year, under the supervision of a dedicated coach specialized in supporting overweighted patients.
  Typical training session organized for small groups (5 patients) will consist of aerobic exercises, muscular strengthening (4 peripheral members and abdominal muscular belt), followed by stretching exercises.
  Arms: Personalized Physical Activity

SUMMARY:
This study compares the ratio of lean mass losses over total body mass losses between patients undergoing sleeve gastrectomy followed by physical activity training versus patients undergoing sleeve gastrectomy only

DETAILED DESCRIPTION:
This study will assess prospectively and objectively the potential benefits of a personalized and specific rehabilitation program designed for patients who undergone sleeve gastrectomy. This strategy will help to reduce fat mass and to limit lean mass loss, in order to prevent in the short term the overweight recurrence. Also,the improvement of physical and metabolic status is expected.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 kg/m² or BMI>35kg/m² with comorbidities qualifying for bariatric surgery
* Stable obesity or obesity evolving for more than 5 years
* Patient cleared by the surgeon for sleeve gastrectomy one month before recruitment
* Absence of contraindication for a sub-maximal stress test
* Performance of a polysomnography before surgery
* Signed informed consent
* Patient benefiting from Health Care Coverage

Exclusion Criteria:

* Absence of preliminary and regular medical check-ups mandatory before sleeve gastrectomy
* Anticipated difficulty for patient follow-up
* Mental diseases (psychosis, depression, suicidal behavior or history)
* Eating disorders
* Lack of informed consent or cooperation
* Unsufficient patient commitment
* Patient under judiciary protection
* Patient not able to comply with any or all the research procedures over time including physical activity
* Patient excluded from the french database of volunteers for clinical trials

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in the ratio of lean mass losses over total body mass losses | 1 month, 6 months, 12 months after surgery
  Percentage of lean mass loss compared to total body weight loss measured with bioimpedancemetry and dual energy X-Rays absorptiometry (DXA) at 1, 6 and 12 months after surgery

SECONDARY OUTCOMES:
Changes in systolic blood pressure | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Change in the Body Mass Index (BMI) | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Anthropometric measures to estimate body Mass Index (BMI).
Changes in the lipid profile | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  (total cholesterol, LDL HDL, Triglycerides)
Changes of glycemia values | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Changes of HbA1C values | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Changes of albuminemia values | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Changes of insulinemia values | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Changes of creatinemia values | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Change in the body composition analysis with segmental analysis | 1 month, 6 months, 12 months after surgery
  Main parameter: Percentage of lean mass loss compared to total body weight loss measured with bioimpedancemetry at at 1, 6 and 12 months after surgery
Change in the qualitative evaluation of physical activity. | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Daily physical activity will be evaluated by a self-questionary (IPAQ)
Change in the quantitative evaluation of physical activity. | 1 month, 6 months and 12 months after surgery
  Daily physical activity will be evaluated by accelerometer measurements.
Sub-maximal stress testing | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
Change in the quantitative evaluation of the sleep quality | Before and 12 months after surgery
  Comparison of sleep quality : micro awakeness index (average number per hour during Rapid Eye Movement (REM) and Non REM phases); index of micro awakeness following an apnea event.
Change in the qualitative evaluation of the sleep quality | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Comparison of the sleep quality by the mean of a visual analogic scale in a sleep diary
Change in the energy balance | 1 month, 6 months, 12 months after surgery
  Energy balance analysis (energy intake vs energy expenditure) and detailed nutriments analysis.
Change in the 6 min Walking test | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Determination of the maximal walking distance performed by the patient after a 6 minutes walk
Change in the quantitative self esteem evaluation | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Rosenberg questionary for the evaluation of Self-esteem
Change in the quantitative evaluation of the health related quality of life | 1 month, 3 months, 6 months, 9 months and 12 months after surgery
  Medical Outcome Study Short Form-36 (MOS SF-36) questionary

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cracco, MD, Principal Investigator — Groupement des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Hopital Saint Philibert, Lomme, France